CLINICAL TRIAL: NCT04160260
Title: A Phase 1 Multi-Center Study to Measure the Pharmacokinetics of Oral Omadacycline in Adult Subjects With Community-Acquired Bacterial Pneumonia (CABP)
Brief Title: Study to Evaluate the PK of PO Omadacycline in Adults With Community-Acquired Bacterial Pneumonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTK0796-CABPPO-19109
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — omadacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omadacycline: Omadacycline Tablets (Experimental)
  Interventions: Drug: Omadacycline

INTERVENTIONS:
Drug: Omadacycline — Omadacycline: PO Tablets
  Other Names: NUZRYA

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of an oral omadacycline dosing regimen in the treatment of adults with CABP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, age 18 or older who have signed the informed consent form
* Must have a qualifying community-acquired bacterial pneumonia
* Has disease severity such that oral antibiotics therapy is appropriate
* Participants must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug
* Must be able to swallow tablets and comply with all of the requirements of the study

Exclusion Criteria:

* Has received more than 24 hours of a potentially effective systemic antibacterial therapy within the 72 hours prior to the first dose of test article
* Known or suspected infection caused by a pathogen that may be resistant to test article
* Participants who reside in a long-term care or nursing home
* Evidence of empyema
* Evidence of significant immunological disease
* Evidence of liver impairment or disease
* Evidence of unstable cardiac disease
* Severe renal disease or requirement for dialysis
* Evidence of septic shock
* Has a history of hypersensitivity or allergic reaction to any tetracycline
* Has received an investigational drug within the past 30 days
* Participants who are pregnant or nursing
* Unable or unwilling to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Site 105, Birmingham, Alabama
  - Site 102, San Diego, California
  - Site 104, San Diego, California
  - Site 111, Clearwater, Florida
  - Site 116, Clearwater, Florida
  - Site 106, Doral, Florida
  - Site 108, Miami, Florida
  - Site 110, Miami, Florida
  - Site 112, West Palm Beach, Florida
  - Site 103, Butte, Montana
  - Site 114, Las Vegas, Nevada
  - Site 101, Sherman, Texas
  - Site 109, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 participants were screened. Of these, 2 participants failed screening, and 18 participants were enrolled in the study.
Groups:
- 300 mg PO Omadacycline: Participants received omadacycline 300 milligrams (mg) per oral (PO) twice daily (BID) on Day 1, followed by omadacycline 300 mg PO once daily (QD) from Day 2 through Day 10.
Period: Overall Study
Arm/Group | 300 mg PO Omadacycline
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All enrolled participants regardless of whether they received the study drug. However, all enrolled participants had received omadacycline during this study.
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Log Geometric Mean Area Under the Concentration Versus Time Curve (AUC) From Time 0 to 48 Hours After Dosing (AUC[0-48]) of Oral Omadacycline on Day 2
Description: AUC(0-48) was calculated using the linear trapezoidal linear interpolation method using WinNonlin validated statistical analysis software (SAS) program. Participants with plasma concentration data above the limit of quantification were included in the analysis for this pharmacokinetic (PK) endpoint. If any participant had an emesis within 4 hours after dosing on Study Days 1 and 2, the participant was excluded from PK Analysis. Data for 100 mg intravenous (IV) omadacycline treatment group which was used for comparison in the statistical analysis were obtained from 6 completed studies: PTK 0796-SDES-0501, PTK 0796-BEQU-0801, PTK 0796 WOIV-0703, CPTK796-A2104, CPTK796-A2201, and PTK 0796-RENL-15102. NCT numbers of these studies were not available.
Time Frame: Day 1: pre-dose; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 13, 13.5, 14, 14.5, 15, 16, and 24 hours post dose. Day 2: pre-dose; 1, 1.5, 2, 2.5, 3, 4, and 6 hours post dose
Population: Pharmacokinetic (PK) Population: All participants who received omadacycline and had at least 1 evaluable PK parameter. Two participants who reported emesis within 4 hours post-dose and 1 participant with only Day 1 PK profile and no sampling on Day 2, were excluded from the analysis in 300 mg omadacycline treatment arm. Two additional participants with unusually low PK concentrations deemed as outliers were excluded from the analysis.
Measure: Geometric Mean (Standard Deviation); unit: Hours x nanograms/milliliter (h*ng/mL)
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 13
Hours x nanograms/milliliter (h*ng/mL) | 9.93 (0.364)
Statistical Analysis 1: Comparison: 300 mg PO Omadacycline; Comparison was performed with the 100 mg intravenous (IV) omadacycline treatment group (data were obtained from 6 completed studies-NCT numbers not available). Using the Day 1 plasma concentration profile of the 100 mg IV QD dosing from these studies, a BID dosing on Day 1 and a QD dosing on Day 2 was simulated using the superposition principle. Log Geometric Mean (GM) AUC(0-48) of omadacycline for the 100 mg IV omadacycline group was as follows:Participants analyzed=63; GM (SD)=9.98 (0.2091); Test type: Equivalence — Omadacycline 300 mg PO provided equivalent total exposure as measured by AUC relative to omadacycline 100 mg IV; Geometric Mean Ratio = 95.17, 90% CI 2-sided [84.2 to 107.5] — A t-test on the natural log-transformed PK parameter AUC(0-48) was performed to obtain the Geometric Mean Ratio and its confidence interval

2. Primary Outcome: Log Geometric Mean AUC From Time 0 to 24 Hours After Dosing (AUC[0-24]) of Oral Omadacycline on Day 1
Description: AUC(0-24) was calculated using the linear trapezoidal linear interpolation method using WinNonlin validated SAS program. Participants with plasma concentration data above the limit of quantification were included in the analysis for this PK endpoint. If any participant had an emesis within 4 hours after dosing on Study Day 1, the participant was excluded from PK Analysis. Data for 100 mg intravenous (IV) omadacycline treatment group which was used for comparison in the statistical analysis were obtained from 6 completed studies: PTK 0796-SDES-0501, PTK 0796-BEQU-0801, PTK 0796 WOIV-0703, CPTK796-A2104, CPTK796-A2201, and PTK 0796-RENL-15102. NCT numbers of these studies were not available.
Time Frame: Day 1: pre-dose; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 13, 13.5, 14, 14.5, 15, 16, and 24 hours post dose
Population: PK population. Two participants who reported emesis within 4 hours post-dose on Day 1 were excluded from the analysis in 300 mg omadacycline treatment arm. Two additional participants with unusually low PK concentrations deemed as outliers were excluded from the analysis.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 14
h*ng/mL | 9.27 (0.502)
Statistical Analysis 1: Comparison: 300 mg PO Omadacycline; Comparison was performed with the 100 mg IV omadacycline treatment group (data were obtained from 6 completed studies-NCT numbers not available). Using the Day 1 plasma concentration profile of the 100 mg IV QD dosing from these studies, a BID dosing on Day 1 and a QD dosing on Day 2 was simulated using the superposition principle. Log GM AUC(0-24) of omadacycline for the 100 mg IV omadacycline group was as follows:Participants analyzed=63; GM (SD)=9.26 (0.1985); Test type: Equivalence — Omadacycline 300 mg PO provided equivalent total exposure as measured by AUC relative to omadacycline 100 mg IV; Geometric Mean Ratio = 100.8, 90% CI 2-sided [88.0 to 115.5] — A t-test on the natural log-transformed PK parameter AUC(0-24) was performed to obtain the Geometric Mean Ratio and its confidence interval

3. Primary Outcome: Geometric Mean AUC From Time 0 to the Last Quantifiable Concentration (AUClast) of Oral Omadacycline on Day 1 and Day 2
Description: AUClast was calculated using the linear trapezoidal linear interpolation method using WinNonlin validated SAS program. Participants with plasma concentration data above the limit of quantification were included in the analysis for this PK endpoint. If any participant had an emesis within 4 hours after dosing on Study Days 1 and 2, the participant was excluded from PK Analysis.
Time Frame: Day 1: pre-dose; 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 13, 13.5,14, 14.5, 15, 16, and 24 hours post dose; Day 2: pre-dose; 1, 1.5, 2,2.5, 3, 4, and 6 hours post dose
Population: PK population. Two participants who reported emesis within 4 hours post-dose were excluded from the analysis. Additionally, 1 participant with only Day 1 PK profile and no sampling on Day 2, was excluded from the Day 2 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
h*ng/mL
  Day 1: number analyzed (Participants) | 16
  Day 1 | 8468.9 (89.9)
  Day 2: number analyzed (Participants) | 15
  Day 2 | 8467.8 (69.9)

4. Primary Outcome: Geometric Mean of Maximum Observed Plasma Concentration (Cmax) of Oral Omadacycline on Day 1 and Day 2
Description: Cmax was calculated using the linear trapezoidal linear interpolation method using WinNonlin validated SAS program. Participants with plasma concentration data above the limit of quantification were included in the analysis for this PK endpoint. If any participant had an emesis within 4 hours after dosing on Study Days 1 and 2, the participant was excluded from PK Analysis.
Time Frame: as for outcome 3
Population: PK population. Two participants who reported emesis within 4 hours post-dose were excluded from the Day 1 analysis. Additionally, 1 participant with only Day 1 PK profile and no sampling on Day 2, was excluded from the Day 2 analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
Nanograms per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 16
  Day 1 | 721.2 (83.9)
  Day 2: number analyzed (Participants) | 15
  Day 2 | 708.6 (68.7)

5. Primary Outcome: Median Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Oral Omadacycline on Day 1 and Day 2
Description: Tmax was calculated using the linear trapezoidal linear interpolation method using WinNonlin validated SAS program. Participants with plasma concentration data above the limit of quantification were included in the analysis for this PK endpoint. If any participant had an emesis within 4 hours after dosing on Study Days 1 and 2, the participant was excluded from PK Analysis.
Time Frame: Day 1: Pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 13, 13.5,14, 14.5, 15, 16, 24 hours post dose; Day 2: Pre-dose, 1, 1.5, 2,2.5, 3, 4, 6 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
Hours
  Day 1: number analyzed (Participants) | 16
  Day 1 | 3.0 [1 to 24]
  Day 2: number analyzed (Participants) | 15
  Day 2 | 2.1 [2 to 3]

6. Primary Outcome: Median Elimination Half-life Associated With the Terminal Slope of the Semilogarithmic Concentration-time Curve (T1/2) of Oral Omadacycline on Day 1 and Day 2
Description: T1/2 was calculated using the linear regression of the terminal portion of the natural log-plasma concentration versus time curve. Participants with plasma concentration data above the limit of quantification were included in the analysis for this PK endpoint. If any participant had an emesis within 4 hours after dosing on Study Days 1 and 2, the participant was excluded from PK Analysis.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 15
Hours
  Day 1 | 8.0 [6 to 16]
  Day 2 | 13.1 [6 to 21]

7. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Treatment-related TEAE, and Serious Adverse Event (SAE)
Description: AEs were defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs were defined as AEs that began (or pre-existing AEs that worsened) on or after the first dose. SAEs were defined as any untoward medical occurrence that, at any dose resulted in: death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may have jeopardized the participant or may have required medical or surgical intervention.
Time Frame: From the first dose of study drug up to 37 days
Population: Safety Population: all enrolled participants who received at least one dose of omadacycline during the study
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
Participants
  TEAEs | 10
  Treatment-related TEAEs | 8
  SAEs | 0

8. Other Pre Specified Outcome: Number of Participants With Clinical Success, Clinical Failure and Indeterminate Clinical Response at the End of Treatment (EOT) as Determined by Investigator Assessment (IGA)
Description: The investigator determined whether or not the participant met the criteria of 1 of the following clinical outcomes: Clinical success, clinical failure, and indeterminate. Clinical success: Participant was alive and the infection was sufficiently resolved such that further antibacterial therapy was not needed. Clinical Failure: Participant required alternative antibacterial treatment for community-acquired bacterial pneumonia (CABP) prior to EOT related to either progression or development of new symptoms of CABP or development of infectious complications of CABP (eg, empyema, lung abscess) or participant developed an AE that required discontinuation of study therapy. Indeterminate: the clinical response to test article could not be adequately inferred.
Time Frame: Up to 37 days
Population: Intent-to-Treat (ITT) Population: All enrolled participants regardless of whether they received the study drug. However, all enrolled participants had received oral omadacycline during this study.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg PO Omadacycline
Number analyzed (Participants) | 18
Participants
  Clinical Success | 18
  Clinical Failure | 0
  Indeterminate | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 37 days
Description: Treatment-emergent adverse events (TEAEs), defined as any AEs that newly appeared, increased in frequency, or worsened in severity on or after the initiation of active test article, were reported for the Safety Population (all enrolled participants who received at least one dose of oral omadacycline during the study).
Arm/Group | 300 mg PO Omadacycline
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 10/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg PO Omadacycline (N=18)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT04160260/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT04160260/SAP_001.pdf